CLINICAL TRIAL: NCT01032317
Title: EZ Steer™ THERMOCOOL® With CF Sensing Capability (THERMOCOOL SMARTTOUCH™) for the Treatment of Atrial Fibrillation and Ventricular Tachycardia
Brief Title: Study of a New Catheter Using Force Sensing Capabilities for the Treatment of Atrial Fibrillation and Ventricular Tachycardia
Acronym: EZCF-125
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZCF-125
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation; Ischemic Ventricular Tachycardia
Keywords: Arrhythmia; Electrophysiology; Fibrillation; Tachycardia; Ablation; Atrial Fibrillation (AF); Ischemic Ventricular Tachycardia (VT)
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Tachycardia | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm Study (Other): This study was completed prior to the implementation of the requirement for specific identification of study arms. As the requirement was not made retroactive to completed studies, we believe this study to be exempt from the stipulation. Also, per PRS definition, since this is for a single-arm/feasibility study, the data elements are optional.
  Interventions: Device: Radiofrequency Catheter Ablation

INTERVENTIONS:
Device: Radiofrequency Catheter Ablation — The Biosense Webster EZ Steer ThermoCool NAV Diagnostic / Ablation Deflectable Tip Catheter with Contact Force Sensing Capability is designed to facilitate electrophysiological mapping and transmit radiofrequency current as well as provide a real-time measurement of contact force.

SUMMARY:
The purpose of this study is to study the treatment of Atrial Fibrillation and ischemic Ventricular Tachycardia using a RF ablation catheter with contact force sensing capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atrial fibrillation or ischemic ventricular tachycardia

Exclusion Criteria:

* Longstanding persistent AF
* Idiopathic VT
* Congestive Heart Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The incidence of early onset (within 7 days of ablation procedure performed with the study devivce) primary adverse events. | 7 days
  The primary safety endpoint is the incidence of early onset primary adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- IKEM, Prague, Czechia